CLINICAL TRIAL: NCT00711087
Title: Botulinum Toxin A Treatment of Detrusor External Sphincter Dyssynergia During Early Spinal Cord Injury (Protocol #H-20344)
Brief Title: Botox-A Injection to Improve Bladder Function in Early Spinal Cord Injury (#H-20344)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funds no longer available
Sponsor: Baylor College of Medicine (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christopher Patrick Smith, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-20344
Record Dates: First submitted 2008-07-07; First posted 2008-07-08 (Estimated); Results first posted 2015-10-09 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Neurogenic Bladder Dysfunction Nos; Spinal Cord Injury
Keywords: Spinal Cord Injury; Bladder; Botulinum toxin (BOTOX-A; Detrusor External Sphincter Dyssynergia
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM 2 (Placebo Comparator): Subjects randomized to receive placebo (saline) sham saline injections on Days 0 and 90.
  Interventions: Other: Saline injection
- ARM 1 (Active Comparator): Subjects randomized to receive 100 units BOTOX-A injections on Days 0 and 90.
  Interventions: Drug: BOTOX-A

INTERVENTIONS:
Drug: BOTOX-A — Group 1-100 units of BTX-A (Botox®, Allergan Inc., Irvine, CA) on Day 0 and 100 units of BTX-A on Day 90
  Other Names: BTX-A; Botulinum Toxin Type A
  Arms: ARM 1
Other: Saline injection — Group 2-sham saline injections on both Day 0 and Day 90.
  Arms: ARM 2

SUMMARY:
The purpose of this study is to see what the effect of Botox has on bladder function for those who have recently suffered spinal cord injury. We also will study bladder tissue levels of NGF (nerve growth factor) that can tell us how the nerves to the bladder are healing after injury.

Consenting male and female cervical and high thoracic (T10 and above) SCI patients will be identified within the first 6-7 weeks after SCI and randomized to two external urethral sphincter injection groups. Each group will be injected within 8 weeks after SCI (Day 0) and 3 months later (Day 90). The injection paradigm will consist of: Group 1-100 units of BTX-A (Botox®, Allergan Inc., Irvine, CA) on Day 0 and 100 units of BTX-A on Day 90; Group 2-sham saline injections on both Day 0 and Day 90. Injections will be performed under local anesthesia using standard flexible cystoscopic equipment.

Use of placebo is justified because: 1. there have been documentation of nerve desensitization with dry needling (i.e. acupuncture) and wet needling (i.e. saline)--therefore, to truly demonstrate benefit of Botox over just the needle insertion into the sphincter muscle or injection of the diluent saline, a sham saline injection group is included, 2. the injection procedure itself is minimally invasive and not expected to result in any complications.

Subjects who qualify and have signed the informed consent document will be randomized into two groups, those receiving the BTX-A and those receiving placebo. Blinding will be performed by the TIRR pharmacy department who will provide Botox and placebo in identical syringes so that the treating staff will be blinded. Pharmacists will ensure patients receive the same agent at the time of the second injection. Unblinding will occur at the end of the study or if complications necessitate breaking of the code. Both groups will undergo urodynamic testing to document before and after treatment data. Bladder biopsies will be taken prior to treatment in both groups that will be analyzed for nerve growth factor. Three day voiding diaries will be kept and reviewed with the study coordinator at the follow up visits. Quality of life questionnaires will be completed at each follow up visit. The treatments will take place on Day 0 and Day 90. Follow up visits will occur at Day 120, 16 month, and 28 months.

DETAILED DESCRIPTION:
Approximately 10,000 spinal cord injuries (SCI) occur each year, most of which occur in males (80%). Many of these patients develop neurogenic bladder dysfunction (NGB) characterized by overactivity of the detrusor muscle, termed detrusor overactivity (DO) or detrusor hyperreflexia (DH). They can also develop detrusor external sphincter dyssynergia (DESD), an abnormal/ uncoordinated response of the sphincter to bladder contraction. A combination of these factors can lead to long-term complications in up to 50% of patients. These complications include hydronephrosis, autonomic dysreflexia, vesicoureteral reflux, nephrolithiasis, sepsis, renal insufficiency or failure and even death. Our basic understanding of the physiology of NGB as well as the introduction of the concept of clean intermittent catheterization (CIC) several decades ago has significantly reduced the death rate due to renal complications in SCI patients. Nevertheless, there continues to be a significant amount of morbidity and risk that these patients experience due to our incomplete understanding of DESD; both its development and subsequent impact on bladder function. We postulate that a primary drive to producing detrusor hypercontractility is the obstruction created by increased tone within the external urethral sphincter (EUS). In addition, we hypothesize that high-pressure obstructive voiding patterns displayed by patients with DESD promote development of bladder wall smooth muscle hypertrophy and fibrosis, loss of bladder compliance, and development of the complications listed above.

Most of our treatment options for neurogenic bladder in the SCI patient population aim to reduce bladder filling pressures and obstructive voiding patterns either by reducing bladder overactivity (i.e. antimuscarinic agents) or by decreasing bladder outlet resistance (i..e. alpha 1-adrenergic receptor antagonists, sphincterotomy, UroLume stent placement, or botulinum toxin injection of external urethral sphincter). However, typically treatments are not initiated until these reflex voiding patterns have already developed. Almost all patients with supraconal lesions, regardless of their neurological level of injury or final voiding patterns, display areflexic bladders during the acute and subacute time period after SCI. This time period can last anywhere from 1 month to 1 year (typically 6-8 weeks) after which spinal reflex voiding develops. Dyssynergic voiding patterns are most common in cervical and thoracic (supraconal) lesions while are flexic voiding patterns predominate in lumbar and sacral conal and infraconal injuries. However, there are many exceptions to this rule, especially in incomplete lesions, and that is why urodynamic testing is an important component in the evaluation of every SCI patient.

Nerve Growth Factor (NGF): Role in Obstructive Uropathy: The processes that lead to reorganization of neural pathways and emergence of hyperactive and dyssynergic voiding are incompletely understood. Possible mechanisms underlying the neural plasticity following SCI could involve alterations in levels of neurotrophic factors within the bladder. Nerve Growth Factor (NGF) is a signaling protein that is thought to play a prominent role in mediating the development of bladder reflex voiding mechanisms in various disorders of bladder dysfunction including neurogenic and non-neurogenic bladder outlet obstruction and chronic bladder inflammation (i.e. interstitial cystitis). Studies have found that by inhibiting NGF's actions through immunization, enhancement of bladder hyperactivity and detrusor sphincter dyssynergia was prevented in SCI rats. Finally, studies in SCI human patients found that bladder hyperactivity as well as bladder NGF tissue levels was significantly reduced by bladder BTX-A treatment.

BOTOX® (Botulinum Toxin Type A) Purified Neurotoxin Complex is a sterile, vacuum-dried purified botulinum toxin type A, produced from fermentation of Hall strain Clostridium botulinum type A grown in a medium containing casein hydrolysate, glucose and yeast extract. It is purified from the culture solution by dialysis and a series of acid precipitations to a complex consisting of the neurotoxin, and several accessory proteins. The complex is dissolved in sterile sodium chloride solution containing Albumin Human and is sterile filtered (0.2 microns) prior to filling and vacuum-drying.

One Unit of BOTOX corresponds to the calculated median intraperitoneal lethal dose (LD50) in mice. The method utilized for performing the assay is specific to Allergan's product, BOTOX®. Due to specific details of this assay such as the vehicle, dilution scheme and laboratory protocols for the various mouse LD50 assays, Units of biological activity of BOTOX cannot be compared to nor converted into Units of any other botulinum toxin or any toxin assessed with any other specific assay method. Therefore, differences in species sensitivities to different botulinum neurotoxin serotypes precludes BOTOX is approximately 20 units/nanogram of neurotoxin protein complex.

Each vial of BOTOX contains 100 Units (U) of Clostridium botulinum type A neurotoxin complex, 0.5 milligrams of Albumin Human, and 0.9 milligrams of sodium chloride in a sterile, vacuum-dried form without a preservative.

Botulinum Toxin (BTX-A) to treat DESD: Botulinum toxin, first isolated by van Ermengem in 1897, is the most potent biological toxin known to man. Through basic and clinical research, clinicians have been able to transform this lethal toxin into a health benefit. BTX-A represents a viable option in the treatment of DESD. When injected, the toxin acts at the neuromuscular junction of the external sphincter to block vesicle transport of acetylcholine; in essence, producing a chemical denervation. The clinical effects begin within 2-3 days and are reversible as terminal nerve sprouting occurs within 3-6 months.

The majority of studies on DESD have examined several outcome measures following BTX-A injection: Change in post-void residual (PVR), change in urethral pressure profile (UPP-static or dynamic), change in bladder pressures during voiding, change in frequency or severity of autonomic dysreflexia (AD), and change in symptoms or satisfaction of the procedure to the patient. Once again, BTX-A treated patients' demonstrated improvements in PVR and UPP similar to their previous study.

However, while most studies of BTX-A for DESD have documented significant reductions in detrusor and urethral pressures as well as PVR, prior research has shown that detrusor leak point pressure (DLPP) is the best prognostic measure for upper tract damage in neurogenic bladder patients. This fundamental concept was corroborated by external sphincterotomy studies demonstrating that failure to achieve a DLPP below 40 cm H2O increases the frequency of upper tract deterioration. This finding underscores the importance that future studies examining the efficacy of BTX treatment for DESD will utilize DLPP as an objective measure of the procedure's success.

Preliminary Data: Effect of BTX-A on Urethral Outlet Resistance by Measuring Changes in Leak Point Pressure. The purpose of these investigations was to evaluate the effects of BTX-A on in vivo urethral resistance by measuring leak point pressure (LPP) with a vertical tilt table and intravesical pressure clamp.

Female SD rats (n=8; 220-250g) were anesthetized with urethane (1.2 g/kg) and injected intraperitoneally with either BTX-A (100u) or saline 18 hours prior to experimentation. LPP was recorded before and after administration of the nicotinic receptor antagonist -bungarotoxin (BGT), and the ganglionic blocker hexamethonium (HEX).

BGT significantly decreased the LPP in control animals by 46% but had no appreciable affect in BTX-A treated animals. In comparison, BTX-A treatment decreased LPP by 47% compared to baseline values in control animals. The ganglionic blocker, HEX, had no appreciable effect on either control or BTX-A treated animals.

BTX-A significantly decreased the basal LPP to the same extent as BGT, confirming it's in vivo potency at the striated neuromuscular junction. However, the fact that HEX had no appreciable effect in either group suggests that sympathetic tone is not a prominent component of outlet resistance in female rats, and may not be a suitable in vivo model to describe the effects of BTX-A on urethral adrenergic pathways. Although originally designed as a method to evaluate stress urinary incontinence in rodents, this method actually measures the intravesical pressure during bladder filling at which urinary leakage occurs, that is, detrusor leak point pressure (DLPP). The marked decrease in DLPP induced by BTX-A in this animal model validates BTX-A's potential effects on DLPP in humans with DESD.

BTX-A Urethral Sphincter Injections in Humans: Sixty eight patients received urethral sphincter injections for bladder outlet obstruction resulting from DESD or pelvic floor spasticity. Patients' mean age was 53 (range 21-71) and the underlying pathophysiology for outlet obstruction included: spinal cord injury (n=9), multiple sclerosis (n=32), stroke (n=4), other (n=8), idiopathic retention/pelvic floor spasticity (n=15). Patients were injected with 100 units of BTX-A into their external urethral sphincters under local or general anesthesia. Postoperatively, significant decreases in maximal detrusor pressures (81cm to 52cm H2O, p<0.05) and post-void residuals (240ml to 88ml, p<0.05) were observed with beneficial effects lasting 3-4 months.

Significance: The significance of these experiments begins with the fact that our proposed intervention occurs during early spinal cord injury (i.e. within 8 weeks) before pathologic bladder reflex pathways have emerged. In addition, our proposed project would be: 1. The largest, prospective randomized trial examining the effects of BTX-A urethral sphincter injection for detrusor external sphincter dyssynergia (DESD) and the first to look at the effect of BTX-A on detrusor leak point pressure (DLPP); 2. The first study to evaluate the role that bladder outlet obstruction by DESD plays in the development of bladder hyperactivity and the development of complications resulting from bladder dysfunction; 3. The first study profiling bladder tissue levels of the signaling protein nerve growth factor (NGF) during early SCI and then again once bladder hyperreflexic patterns develop, and; 4. The first study evaluating the effect of reducing outlet resistance with BTX-A on bladder NGF levels. If our hypotheses prove to be correct, treated patients will display less incontinence, require lower doses of anticholinergic medication, and avoid the complications of DESD listed earlier in this proposal. Although this study as written is of moderate length (i.e. total 5 years), we hope that by finding significant results we will be able to capture a longitudinal history of this population by extending follow-up to a longer duration (i.e. >10 years). In addition, BTX-A treatment could be extended to other neurogenic populations suffering from DESD (i.e. Multiple Sclerosis) as well as other conditions where bladder overactivity appears to be driven by outlet obstruction (i.e. Benign Prostatic Hyperplasia).

Hypotheses:

1. BTX-A injection of the external urethral sphincter significantly decreases detrusor leak point pressure (DLPP).
2. Decreased DLPP during early SCI will markedly reduce bladder tissue nerve growth factor (NGF).
3. Reducing DLPP and bladder NGF during early SCI will diminish complications associated with neurogenic detrusor overactivity (NDO) and outlet obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Male or Females between ages of 18-50
* Patient weighs over 111 pounds
* Patient has documented Spinal Cord Injury T10 or above Thoracic Level by ASIA Score less than 8 weeks prior to the start of the study. Both complete and incomplete spinal cord injuries will be included in this study.
* Ability to complete all study requirements including voiding diary and to attend all scheduled study visits, in the opinion of the investigator
* Written informed consent has been obtained
* Patient has negative pregnancy test result if female and of child-bearing potential
* Written authorization for use and release of Health and Research Study Information has been obtained
* Patient or family member is willing and able to perform clean intermittent catheterization for duration of this study

Exclusion Criteria:

* Patient has received anticholinergic medication for the treatment of overactive bladder before randomization into the study
* Patient has history or evidence of any pelvic or urological abnormalities, bladder or urethral surgery or disease, other than neurogenic bladder related to spinal cord injury, that may impact bladder function
* Patient has significant stress urinary incontinence, determined by patient history, in the opinion of the investigator
* Neurogenic detrusor overactivity (greater than 10cm elevation in pdet pressure) at baseline urodynamic screening (Day 0)
* Patient found to have significant baseline renal pathology (e.g. hydronephrosis, stones, renal mass) at Day -7
* Patient has a history of two or more treated urinary tract infections within 6 months of screening Day -7
* Patient has urinary tract infection defined as a bacteriuria count of greater than 105/ml conjoint with leukocyturia greater than 5hpf at screening Day -7
* Patient has asymptomatic urinary tract infection, defined as positive nitrites, leukocyte esterase and or blood on urine dipstick reagent strip at randomization Day 0
* Patient has history of unexplained hematuria or unexplained hematuria if greater than 5 RBC's/hpf are present at screening Day -7
* Patient has active genital infection, other than genital warts, either concurrently or within 4 weeks prior to screening Day -7
* Patient has history of interstitial cystitis, in the opinion of the investigator
* Patient has evidence of urethral obstruction, in the opinion of the investigator at screening Day -7 or randomization Day 0
* Patient uses medications with anti-platelet or anti-coagulant effects (except Lovenox) within 10 days of randomization Day 0. Lovenox 30mg SQ every 12 hours is standard of care after SCI until 2-3 months post injury. Lovenox will be stopped 24 hours before and for 48 hours after each sphincter injection or bladder biopsy procedure.
* Patient has hemophilia, or other clotting factor deficiencies or disorders that cause bleeding diathesis
* Patient has previously been treated with any endovesical pharmacologic agent (e.g. capsaicin, resiniferatoxin)
* Patient has had previous or current botulinum toxin therapy of any serotype for any condition
* Patient has a known allergy or sensitivity to any components of the study medication, anesthetics or antibiotics to be used during the study
* Any medical condition that may put the patient at increased risk with exposure to Botox® including diagnosed myasthenia gravis, Eaton-Lambert syndrome or amyotrophic lateral sclerosis
* Females who are pregnant, nursing or planning a pregnancy during the study or females of child-bearing potential who are unable or unwilling to use a reliable form of contraception during the study
* Current or previous participation in another therapeutic study within 30 days of screening Day -7
* Any condition or situation which, in the investigator's opinion, puts the patient at significant risk, could confound the study results, or may interfere significantly with the patient's participation in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2007-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P. Smith, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Memorial Hermann Hospital/The Institute of Rehabilitation and Research, Houston, Texas

REFERENCES:
- [Background] Smith CP, Chancellor MB. Emerging role of botulinum toxin in the management of voiding dysfunction. J Urol. 2004 Jun;171(6 Pt 1):2128-37. doi: 10.1097/01.ju.0000127725.48479.89. PMID 15126771
- [Background] Smith CP, Nishiguchi J, O'Leary M, Yoshimura N, Chancellor MB. Single-institution experience in 110 patients with botulinum toxin A injection into bladder or urethra. Urology. 2005 Jan;65(1):37-41. doi: 10.1016/j.urology.2004.08.016. PMID 15667859

RESULTS

PARTICIPANT FLOW:
Groups:
- ARM 2: Patients in ARM 2 randomized to receive placebo (saline) injections on Days 0 and 90.
- ARM 1: Patients in ARM 1 randomized to receive 100 units of BOTOX-A on Day 0 and Day 90
Period: Overall Study
Arm/Group | ARM 2 | ARM 1
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only one (1) patient was enrolled on this study. That participant was randomized to Arm 1.
Groups:
- ARM 1: Subjects randomized to this group will receive placebo.
- ARM 2: Subjects randomized to receive 100 units of BOTOX-A injections on Days 0 and 90.
- Total: Total of all reporting groups
Arm/Group | ARM 1 | ARM 2 | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] |  | 1 [0 to 100] | 1 [0 to 100]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: A Change in DLPP of 20cm H2O at Day 30 and Day 120 in the BTX-A Injected Group (Group 1) Compared to the Sham Saline Injected Group (Group 2).
Description: This outcome measure was not able to be determined due to the subject being lost to follow-up. The subject no longer returns phone calls or visits the clinic.
Time Frame: 2.5 years
Population: Early spinal cord injury
Groups:
- ARM 1: Subjects randomized to receive 100 units of BOTOX-A on Days 0 and 90
Arm/Group | ARM 2 | ARM 1
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse events were collected over a period of 28 months.
Description: Unreported major toxicity (Grade 4 or 5). Repetitive failure to report Grade 2 - 3 toxicities. Serious or repetitive failure to properly characterize toxicity or grade. Failure to file required NCI Adverse Event Reports according to the protocol and NCI Guidelines if applicable.
  There was one patient enrolled and that patient did not have any adverse or serious adverse events.
Groups:
- ARM 2: Receiving placebo (saline injections)
  Saline injection: Group 2-sham saline injections on both Day 0 and Day 90.
- ARM 1: Receiving BOTOX-A
  BOTOX-A: Group 1-100 units of BTX-A (Botox®, Allergan Inc., Irvine, CA) on Day 0 and 100 units of BTX-A on Day 90
Arm/Group | ARM 2 | ARM 1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No